CLINICAL TRIAL: NCT04928157
Title: Prospective Randomized Trial of CPAP for SDB in Patients Who Use Opioids
Acronym: PRESTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeremy Orr, M.D., Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201743; K23HL151880 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Sleep Disorder; Breathing-Related; Pain; Sleep Apnea; Obstructive Sleep Apnea; Sleep; Sleep Disorder; Chronic Pain; Opioid Use
Keywords: sleep; sleep apnea; OSA
MeSH Terms: conditions — Sleep Wake Disorders; Pain; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CPAP (Experimental): Use of CPAP, a device used with a nose or face mask which delivers airflow/pressure into the airway, holding the airway open and keeping it from collapsing. Device will be used for 8 weeks.
  Interventions: Device: Positive Airway Pressure (PAP)
- Control (No Intervention): No CPAP use, otherwise usual care

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) — A device used with a nose or face mask which delivers airflow/pressure into the airway, holding the airway open and keeping it from collapsing. Device will be used for 8 weeks.
  Other Names: CPAP
  Arms: CPAP

SUMMARY:
Patients with chronic pain who use opioids appear to be at increased risk for breathing issues during sleep, termed sleep disordered breathing (SDB). Treatment of SDB often consists of use of a device during sleep that provides continuous positive airway pressure (CPAP) via a mask interface. The goal of this study is to determine whether patients with chronic pain who use opioids and have SDB might benefit from the use of CPAP in terms of sleep quality, pain, quality of life, and other measures. In addition, the study will examine whether these individuals are able to adhere to CPAP, which will be important for future studies. Lastly, we anticipate that CPAP won't work for everyone due to the changes that opioids can cause in breathing patterns. We will examine how often CPAP is ineffective, and whether we can predict which individuals are least likely to resolve their SDB with CPAP.

DETAILED DESCRIPTION:
Patients who use chronic opioids for chronic pain daily for >3 months will be recruited. Patients with recently diagnosed sleep disordered breathing (SDB; defined as an apnea-hypopnea index >/=5 events/hr) will be studied, but a screening sleep study can be performed if the participant has not had a sleep study, and they will be included if SDB is found. Persons who are already under treatment for SDB with continuous positive airway pressure (CPAP) will be excluded, along with those with, recreational opioid use, cancer pain, limited life expectancy, prisoners, pregnant women, psychiatric disease, and those unable to provide consent or cooperate with research procedures. Potential subjects will discuss the planned research protocol, risks, benefits, and alternatives with the study staff.

Once the individual has given written informed consent, they will be scheduled for a baseline study visit, which will begin in the early evening. Subjects will undergo a comprehensive history and physical exam, questionnaires examining sleep quality, daytime function, pain, and quality of life. The cold pressor test will be administered, which includes submerging the non-dominant hand in a 4 degree Celsius water bath, and reporting the onset of pain and maximal tolerable submersion time.

After these procedures, the subject will be instrumented for an overnight sleep study, which will include the application of electrodes to the scalp (electroencephalogram), beside the eyes (electro-oculogram), chin and legs (electromyogram). Elastic bands will be applied around the chest and abdomen, a pulse oximeter will be affixed to the finger, and airflow monitors placed just inside the nose and outside the mouth. The subject will then be allowed to sleep until the morning. Upon awakening, they will undergo a computer test of alertness.

The subject will then be randomized to two groups. One group will be randomized to active CPAP treatment, for which they will be fitted with a nasal mask and instructed on the use of a commercial self-titrating CPAP machine. They will wear the device each night for the next 8 weeks. Use of the device will be monitored by the study staff, and the subject will be contacted by telephone on a weekly basis to address any issues. The other group will be randomized to usual care, which does not include CPAP treatment during this 8 week time interval.

After 8 weeks, subjects will return to the laboratory and undergo the same testing as the baseline visit. For the sleep study, those in the CPAP group will wear their CPAP device during the recording, while the other group will be tested without CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Chronic pain
* Chronic opioid use (daily use for >3 months duration)
* Apnea-hypopnea index >/= 5 events/hr (screening sleep study will be performed)

Exclusion Criteria:

* Already using CPAP or non-invasive ventilation on a daily basis
* Use of opioids outside medical supervision (i.e. recreational use)
* Pain due to active cancer
* Prisoners
* Pregnancy
* Psychiatric illness other than treated mood disorders
* Life expectancy <12 months
* Anticipated inability to sleep in the laboratory setting or to use CPAP
* Unable or unwilling to provide informed consent or comply with research procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
PROMIS sleep disturbance | 8 weeks
  A questionnaire to assess self-reported quality of general sleep and sleep disturbance. Each item on the form is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.

SECONDARY OUTCOMES:
Brief pain inventory | 8 weeks
  Pain questionnaire

OTHER OUTCOMES:
Pain 11 point Likert scale | 8 weeks
  Subjects will be asked to rank their "current pain level" on a scale of 0-10, where 0 is no pain and 10 is the worst possible pain.
Insomnia Severity Index (ISI) | 8 weeks
  A 7-item self-report form to assess insomnia severity. Total score categories: 0-7 = No clinically significant insomnia, 8-14 = Subthreshold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe).
PROMIS Sleep-Related Impairment (SRI) | 8 weeks
  Self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness.
Epworth Sleepiness Scale (ESS) | 8 weeks
  A self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Current Opioid Misuse Measure (COMM) | 8 weeks
  A brief patient self-assessment to monitor chronic pain patients on opioid therapy.
Pittsburg Sleep Quality Index (PSQI) | 8 weeks
  A 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Neuropathic pain scale short form | 8 weeks
  A brief patient self-assessment to measure neuropathic pain symptoms, as well as assisting in discrimination between neuropathic and non-neuropathic pain.
Beck Depression Inventory | 8 weeks
  he questionnaire assesses mental health (i.e. depression). Each of the 21 items are given weighted values corresponding to a symptom of depression and summed to give a single score. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Psychomotor Vigilance (PVT) | 8 weeks
  A 10-minutes, computerized reaction test asking subject to press a button every time a prompt appears. Faster times indicate better reactions and higher alertness.
Apnea Hypopnea Index | 8 weeks
  The number of times a person stops breathing and periods of shallow breathing with a marked decrease in blood oxygen concentration every hour on average. A score lower than five indicates normal sleep (no sleep apnea), 5-15 indicates mild sleep apnea, 15-30 indicates moderate sleep apnea, and a score greater than 30 indicates severe sleep apnea.
Cold Pressor Test | 8 weeks
  The cold pressor test will be performed to assess pain threshold and tolerance. Participants will immerse their hand into a cold water bath, and will be instructed to report the first painful sensation after immersion. They will then be asked to tolerate the stimulus as long as possible, but will be permitted to withdraw their hand from the cold water at any point. Maximum immersion time will be 5 mins. Latency to first feel pain (pain sensitivity) and latency to withdraw the hand from the water (pain tolerance) will be recorded. Blood pressure and heart rate will be measured before and after each immersion using the arm that was not immersed in the water bath.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Orr, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared with other qualified investigators with local IRB approval
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Orr JE, Bosompra NO, Norby B, Velazquez J, Khalaf A, DeYoung P, Schmickl CN, Sands SA, Jain S, He F, Goodin B, Wallace M, Owens RL, Malhotra A. Chronic pain is associated with sleep apnea severity but attenuated by intermittent hypoxemia in people using opioids. Pain. 2026 Jan 1;167(1):159-167. doi: 10.1097/j.pain.0000000000003760. Epub 2025 Jul 24. PMID 40705710
- See also: UCSD Sleep Research Website — http://sleepresearch.ucsd.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04928157/ICF_000.pdf